CLINICAL TRIAL: NCT04259970
Title: Hyperpolarized Imaging for New Treatments (HyPOINT) Study
Brief Title: Hyperpolarized Imaging for New Treatments
Acronym: HyPOINT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Virginia (Other); University of Wisconsin, Madison (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2019-1051
Record Dates: First submitted 2020-01-15; First posted 2020-02-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CFTR modulator therapy; 129Xe MRI; hyperpolarized xenon; LCI
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Phase 1 will include implementation of a centralized analysis program of repeated 129Xe MRI scanning in CF patients with mild lung disease to define the intra-subject variability of the primary outcome ventilation defect percentage (VDP). Patients will undergo baseline 129Xe MRI scanning and repeated measurements the same day, as well as at 28 days (± 7 days). Phase 1 will establish the intra-subject reproducibility to facilitate future use of 129Xe MRI in multi-site studies. Furthermore, the reproducibility limits defined will inform the overall design of future studies and will compare to established pulmonary function and multiple-breath washout testing (via measurement of the lung clearance index, LCI).
  Interventions: Drug: Initiation of CFTR Modulator
- Initiation of CFTR Modulator (Experimental): Phase 2 will be an observational study of patients assessed before and after the clinical initiation of triple-combination modulator therapy (after presumed FDA and Health Canada approval). The primary endpoint for Phase 2 is the change of VDP after 28 days of triple-combination modulator therapy. Within Phase 2, this study will also address how highly-effective modulator therapies affect lung function trajectories by measuring 129Xe MRI at 28 days (± 7 days), 6 months (± 28 days), and 12 months (± 28 days) after start of therapy (paralleling time points of the PROMISE study). Finally, to understand how 129Xe MRI can be used in combination with existing measures of lung function (e.g. spirometry, multiple breath washout), the investigators will directly compare the repeated data collected in both Phase 1 and Phase 2 to these established measures of lung function that are currently used in observational and interventional studies.
  Interventions: Drug: Initiation of CFTR Modulator

INTERVENTIONS:
Drug: Initiation of CFTR Modulator — Inhaled contrast for MRI occurring at each 4 visits.
  Other Names: 129Xe

SUMMARY:
The introduction of triple combination CFTR modulator therapy for patients with Cystic Fibrosis (CF) with at least one copy of the deltaF508 mutation is expected to provide major health benefits, but will also require novel outcome measures that can detect CF lung disease at an early stage, capture the efficacy of new therapies when disease manifestations are limited, as well as determine whether stopping existing chronic maintenance therapies does not have negative effects.

In the past decade, research has focused on the multiple breath washout (MBW) test, as a sensitive outcome measure, especially if highly-effective modulator therapies are initiated in early childhood. Even LCI, however, may not adequately capture early lung function changes, thus warranting investigation of even more sensitive outcome measures.

Magnetic resonance imaging (MRI) has the advantage of being a radiation-free modality, making it more suitable for assessing response to therapy in a shorter time frame with repeated imaging. Inhalation of a hyperpolarized gas enables the visualization and quantification of regional ventilation in the lung and can be combined with structural MRI to assess both structure and function in parallel.

The main Investigator and others have recently formed an international consortium (the 129Xe MRI Clinical Trial Consortium), comprised of both imaging experts and pulmonary clinicians to standardize imaging procedures, thus facilitating multi-site implementations. Data from this proposed study (HyPOINT; Hyperpolarized Imaging for New Treatments) will inform the future utility of MRI for both longitudinal studies to track disease progression over time as well as for future interventional trials. Further, the current study could inform the design of future trials of interventions of patients for whom currently no effective CFTR modulator therapy is available and for patients with rare genotypes thus laying the groundwork for a more personalized medicine approach in the near-term future.

DETAILED DESCRIPTION:
The HyPOINT (HyperPOlarized Imaging for New Therapies) trial is a multicenter prospective, two phase study involving four sites with proven expertise 129Xe MRI and CF clinical care. The study sites are: University of Virginia, University of Wisconsin, and SickKids in Toronto, Canada. University of Virginia and University of Wisconsin sites will be reliant on CCHMC's IRB. SickKids in Toronto, Canada, will submit their review through their institution's Research Ethics Board (REB).

Phase 1 will include implementation of a centralized analysis program of repeated 129Xe MRI scanning in CF patients with mild lung disease to define the intra-subject variability of the primary outcome ventilation defect percentage (VDP). Patients will undergo baseline 129Xe MRI scanning and repeated measurements the same day, as well as at 28 days (± 7 days). Phase 1 will establish the intra-subject reproducibility to facilitate future use of 129Xe MRI in multi-site studies. Furthermore, the reproducibility limits defined will inform the overall design of future studies and will compare to established pulmonary function and multiple-breath washout testing (via measurement of the lung clearance index, LCI).

Safety of 129Xe MRI will be assessed by recording adverse events during the study visit (see 8.3 Adverse Events and Serious Adverse Events), which will be followed until resolved. Vital signs (heart rate, SPO2) will be recorded before, immediately following inhalation, and 2 minutes after each 129Xe inhalation; O2 saturation will be monitored continuously throughout the 129Xe portion of the MRI, and the time and duration of nadir will be recorded.

Phase 2 will be an observational study of patients assessed before and after the clinical initiation of triple-combination modulator therapy (after presumed FDA and Health Canada approval). The primary endpoint for Phase 2 is the change of VDP after 28 days of triple-combination modulator therapy. Within Phase 2, this study will also address how highly-effective modulator therapies affect lung function trajectories by measuring 129Xe MRI at 28 days (± 7 days), 6 months (± 28 days), and 12 months (± 28 days) after start of therapy (paralleling time points of the PROMISE study). Finally, to understand how 129Xe MRI can be used in combination with existing measures of lung function (e.g. spirometry, multiple breath washout), Investigators will directly compare the repeated data collected in both Phase 1 and Phase 2 to these established measures of lung function that are currently used in observational and interventional studies.

The overarching goal of this study is to define the role of structural and functional MRI imaging to facilitate future CF research studies.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative.
2. Willingness and ability to adhere to the study visit schedule and other protocol requirements.
3. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   1. Sweat chloride equal to or greater than 60 mEq/liter by quantitative pilocarpine iontophoresis test
   2. Two well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
4. Phase 1 only: Age 6 to 18 years, inclusive, at the time of consent.
5. Phase 2 only: Ages 9 to 18 years, inclusive, at the time of consent.
6. Clinically stable with no acute antibiotic usage in the 14 days prior to the first visit.
7. Genotype with F508del on at least one allele.
8. No change in chronic pulmonary medications or therapies in the 28 days prior to the first visit.
9. Stable CFTR modulator therapy (TEZ/IVA or LUM/IVA) for at least 28 days prior to the first visit or currently not receiving CFTR modulator therapy.
10. Ability to cooperate with MRI procedures.
11. Phase 1 only: FEV1 greater than or equal to 80% predicted based on GLI reference equations.

Exclusion Criteria:

1. Standard MRI exclusions (Metal implants, claustrophobia).
2. For females of childbearing potential: Positive urine pregnancy test at Screening or Visit 1 or Lactating.
3. Any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Xe VDP Assessment | 28 days
  The primary analysis will use a paired, non-parametric test (e.g., Wilcoxson Rank sum) to determine if the change in VDP from baseline to 28 days is statistically different from no change in VDP.
The change in Xe VDP after 28 days of triple modulator CFTR therapy | 28 days
  To understand how triple combination therapy affects lung function in the long term, we will compare the changes in VDP (summarized as the average change from baseline at 6 months and 12 months), using the same non-parametric matched analysis. This will inform the natural history of VDP and whether future studies of hyperpolarized 129Xe MRI should be designed to show an improvement in VDP or maintenance of VDP. Exploratory analyses using a mixed-effects regression model will be done to define the rate of change of VDP over the 12-month study period.

SECONDARY OUTCOMES:
Overall UTE MRI reader score analysis | 28 days
  The primary analysis will use a paired, non-parametric test (e.g., Wilcoxson Rank sum) to determine if the change in VDP from baseline to 28 days is statistically different from no change in VDP.
The change in overall MRI reader score for UTE MRI 28 days after triple combination therapy is initiated | 28 days
  To understand how triple combination therapy affects lung function in the long term, we will compare the changes in VDP (summarized as the average change from baseline at 6 months and 12 months), using the same non-parametric matched analysis. This will inform the natural history of VDP and whether future studies of hyperpolarized 129Xe MRI should be designed to show an improvement in VDP or maintenance of VDP. Exploratory analyses using a mixed-effects regression model will be done to define the rate of change of VDP over the 12-month study period.
Fev1 and LCI Correlation | 28 days
  A Spearman correlation will be used to determine the correlation between VDP and LCI at each study time points. A similar correlation analysis will be repeated for the change in LCI from baseline and change in VDP from baseline at each of the study time-points. With the treatment data, we will determine the concordance between the two outcomes at detecting an improvement in lung function and investigate where the two tests are discordant. A receiver operator characteristic curve will compare the diagnostic accuracy of the 129Xe MRI, and LCI. Similar analysis will be performed comparing VDP to the FEV1 and comparing the UTE MRI reader score to both LCI and FEV1. Secondary analysis will compare these changes in PFTs and LCI to changes in UTE MRI reader score and to sub-categories of regional ventilation using 129Xe MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
- The Hospital for Sick Kids, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wielputz MO, Puderbach M, Kopp-Schneider A, Stahl M, Fritzsching E, Sommerburg O, Ley S, Sumkauskaite M, Biederer J, Kauczor HU, Eichinger M, Mall MA. Magnetic resonance imaging detects changes in structure and perfusion, and response to therapy in early cystic fibrosis lung disease. Am J Respir Crit Care Med. 2014 Apr 15;189(8):956-65. doi: 10.1164/rccm.201309-1659OC. PMID 24564281